CLINICAL TRIAL: NCT03917043
Title: A Phase I Study of the Safety, Pharmacokinetic and Pharmacodynamic Properties of Orally Administered APG-2449 in Patients With Advanced Solid Tumors
Brief Title: APG-2449 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG2449XC101
Record Dates: First submitted 2019-03-25; First posted 2019-04-16 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Cancer; Non Small Cell Lung Cancer; Esophageal Cancer; Ovarian Cancer; Malignant Pleural Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Ovarian Neoplasms; Mesothelioma, Malignant

STUDY DESIGN:
Intervention Model Description: Dose escalation of APG-2449 will use standard 3+3 design. The starting dose is 150 mg and will be increased in subsequent cohorts to 300mg, 450mg, 600mg, 750mg, 900mg, 1200mg and 1500mg, accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- APG-2449 (Experimental): APG-2449 will be explored sequentially using a standard 3+3 escalation scheme at the dose escalation phase and up to 30-40 patient at the MTD/RP2D dose level.
  Interventions: Drug: APG-2449

INTERVENTIONS:
Drug: APG-2449 — Capsule, multiple dose cohorts, oral administration every day (QD) of a 28-day cycle
  Other Names: APG-2449 Capsule

SUMMARY:
APG-2449 is a novel, orally active, multi-targeted tyrosine kinase inhibitor, which inhibits FAK, ALK, and ROS1 with nanomolar potencies. In preclinical studies, APG-2449 demonstrated potent antiproliferative activity in various cancer cell lines as a single agent. In combination treatment, APG-2449 enhanced anti-proliferative activities of several chemotherapeutic and targeted agents. It is indicated that APG-2449 may have a broad therapeutic potential for the treatment of human cancer as a single agent and in combination with other classes of anticancer drugs. APG-2449 is intended for the treatment of patients with advanced solid tumors. Upon completion of the Phase 1 dose escalation study to establish the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and/or recommended phase 2 dose (RP2D), several phase Ib/II studies will be implemented accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Dose exploration stage: non-small cell lung cancer diagnosed by histology and/or cytology and positive for ALK/ROS1 gene fusion (molecular diagnosis confirmed by the investigator) and malignant pleural mesothelioma, esophageal cancer and ovarian cancer. Kind of patients with advanced tumors.

   Expansion stage: cohort 1, patients with non-small cell lung cancer who have progressed or are intolerant to TKI therapy, including patients with second-generation ALK TKI, or either ROS1 TKI, or third-generation ALK inhibitor (lorlatinib, etc.) with pFAK expression (pFAK expression is subject to central laboratory results) of about 10 or above; Cohort 2, TKI-naïve patients with ALK/ROS1 fusion gene positive NSCLC. The molecular diagnosis results of the above patients can be confirmed by the investigator.
2. ECOG Performance Status ≤ 1.
3. Expectation of life ≥ 3 months.
4. According to RECIST version 1.1, there is at least 1 measurable lesion.
5. Adequate hematologic and bone marrow functions.
6. Adequate renal and liver function.
7. Normal cardiac function.
8. Brain metastases with clinically controlled neurologic symptoms.
9. Serum pregnancy test results of women of childbearing age were negative within 7 days before taking the first dose of study drug.
10. Men, women of childbearing age (postmenopausal women must have been menopausal for at least 12 months before they can be considered infertile) and their partners voluntarily take the study drug for at least 30 days after signing the informed consent form and taking the study drug as deemed effective by the investigator Contraceptive measures
11. Ability to understand and willingness to sign a written informed consent form
12. Subjects must be willing and able to complete the research procedures and follow-up inspections.
13. Subjects are required to provide fresh (for recurrent subjects only) or archived tumor tissue samples from within 28 days prior to treatment. If none of these specimens are available, they may be included after consultation with the sponsor.
14. Subjects should provide fresh biopsy tumor tissue specimens prior to treatment.

Exclusion Criteria:

1. Receiving concurrent anti-cancer therapy (chemotherapy, radiotherapy, immunotherapy, biologic therapy); or any investigational therapy within 28 days prior to the first dose of study drug.
2. Receiving TKI therapy within 8 days prior to the first dose of study drug.
3. Continuance of toxicities due to prior therapy that do not recover (CTCAE V5.0 Grade> 1).
4. Has difficulty in swallowing, absorbing barrier, or other diseases blocking APG-2449' taken.
5. Obvious cardiovascular disease history.
6. Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry.
7. Active symptomatic fungal, bacterial and/or viral infection including, but not limited to, active human immunodeficiency virus (HIV) or viral hepatitis (B or C).
8. Known allergies to study drug ingredients or their analogs.
9. Female subjects who are pregnant or breastfeeding, or expecting to become pregnant during the study period.
10. According to the judgment of the investigator or sponsor, any symptoms or disease of the subject may endanger its safety or interfere with the safety assessment of the study drug.
11. Subjects who have used CYP3A4, CYP2C9, or CYP2C19 moderately potent inhibitors or moderately potent inducers 1 week before receiving the study drug for the first time.
12. Subjects who used CYP3A4 substrates and narrow treatment window 1 week before the first study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  To determine the maximum tolerated dose (MTD) of APG-2449 in subjects with advanced solid tumors
Recommended Phase 2 dose (RP2D) | 28 days
  To determine the tentative recommended Phase 2 dose (RP2D) of APG-2449 in subjects with advanced solid tumors

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 days
  Maximum plasma concentration (Cmax) will be assessed on all participants with APG-2449 treatments
Area under the plasma concentration versus time curve (AUC) | 28 days
  Area under the plasma concentration versus time curve (AUC) will be assessed on all participants with APG-2449 treatments
Phosphorylation of FAK protein | 28 days
  Phosphorylation of FAK protein will be assessed in peripheral blood mononuclear cells on all participants with APG-2449 treatments
Preliminary efficacy assessment: Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 | 4 weeks
  To assess preliminary efficacy in subjects with solid tumors using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Professor, Principal Investigator — Sun Yat-sen University
Locations (9):
- China (9):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun-Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The First affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Provincial Oncology Hospital, Zhengzhou, Henan
  - Union Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Provincial Oncology Hospital, Changsha, Hunan
  - Zhejiang Provincial Oncology Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Ma Y, Song Z, Chen J, Zhao Y, Fang W, Guo Y, Dong Y, Yang Y, Wu G, Fang J, Lin X, Li J, Huang Y, Zhao Y, Hong S, Xue J, Zhang Y, Liu Q, Yang C, Xu L, Yang Y, Xiong D, Yang D, Zhai Y, Zhang L, Zhao H. Safety, pharmacokinetic, pharmacodynamic, and efficacy properties of orally administered APG-2449 in patients with advanced ALK + and ROS1 + non-small-cell lung cancer: a multicentre, open-label, single-arm phase 1 trial. EClinicalMedicine. 2025 Oct 16;89:103556. doi: 10.1016/j.eclinm.2025.103556. eCollection 2025 Nov. PMID 41146927
- [Derived] Fang DD, Tao R, Wang G, Li Y, Zhang K, Xu C, Zhai G, Wang Q, Wang J, Tang C, Min P, Xiong D, Chen J, Wang S, Yang D, Zhai Y. Discovery of a novel ALK/ROS1/FAK inhibitor, APG-2449, in preclinical non-small cell lung cancer and ovarian cancer models. BMC Cancer. 2022 Jul 11;22(1):752. doi: 10.1186/s12885-022-09799-4. PMID 35820889